CLINICAL TRIAL: NCT03957538
Title: The Effect of a VIrtual RealiTy Immersive Experience Upon Anxiety Levels in Patients Undergoing CArdiac caTHeterisation: The VIRTUAL CATH Trial
Brief Title: UHW Angiogram Video Project
Acronym: VIRTUAL CATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Wales (Other)
Responsible Party: Principal Investigator, Holly Morgan, Cardiology Spr, University Hospital of Wales
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17/DEC/7157
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard consent and explanation
- Virtual reality (Experimental): Addition of VR headset
  Interventions: Behavioral: Virtual reality angiogram experience video

INTERVENTIONS:
Behavioral: Virtual reality angiogram experience video — The VR video is watched via the VR headset, and describes the pre- procedural and procedural experience. Concurrent audio will be provided through earplugs to compete the patients' immersive experience. The video was written and directed by the team, and care has been taken to ensure that the same procedural information is contained within both the British Heart Foundation cardiac catheterisation video and of VR immersive video. Filming was performed within the cardiac catheterisation labs at our tertiary centre using the professional services of Orchard Media (Cardiff, UK). The investigators utilized real physicians and nurses to re-enact a typical day for a mock patient undergoing an uncomplicated procedure. There is also a short explanation of the procedure and animations explaining technical aspects of the procedure contained within the VR video.
  Arms: Virtual reality

SUMMARY:
This study is a randomised control trial which aims to assess whether the use of an immersive virtual reality angiogram experience decreases peri-procedural anxiety in patients undergoing cardiac catheterisation.

DETAILED DESCRIPTION:
Patients undergoing cardiac catheterisation are understandably anxious. This is due to a lack of familiarity with both the hospital environment and the planned procedure. Anxiety may negatively affect their patient experience. Appropriate patient information can help improve understanding and reduce anxiety. In particular, video-based patient information prior to cardiac catheterisation has been shown to improve patient's knowledge and reduce peri-procedural anxiety. Generic video-based patient information about the cardiac catheterisation procedure is widely available. Ideally any patient information delivered pre-cardiac catheterization would be specific to the hospital delivering care. The use of virtual reality (VR) in healthcare is novel, but expanding rapidly. The immersive nature of VR allows patients a unique opportunity to prepare for the procedure and environment within which they will be treated. To date, the use of VR to prepare patients for invasive cardiac procedures has not been studied.

The aim of this study is to assess whether the use of an immersive VR experience decreases peri-procedural anxiety in patients undergoing cardiac catheterisation. The investigators will also assess whether the VR experience improves overall patient satisfaction.

With the help of a local media company, a VR cardiac catheterisation video was produced (Figure 1 depicts a screenshot from the VR video). The video is watched with a VR headset to create a 360 immersive experience. The investigators are undertaking a single-centre randomised control trial comparing the use of an immersive VR experience 1 week prior to catheterisation with standard pre-procedural care. Pre procedural anxiety levels and procedural knowledge are assessed by questionnaire, using the validated six-item short-form of the Strait Trait Anxiety Inventory (STAI). A satisfaction questionnaire is also completed before the patient is discharged.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing their first cardiac catheterisation

Exclusion Criteria:

* Patients who cannot comprehend English or Welsh
* Those who have significant visual or auditory impairment meaning they would be unable to fully appreciate the video material

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Difference in pre and post procedural anxiety scores between patients receiving standard care and those who experienced the immersive VR experience | 3 months
  Study data collection will be via questionnaire, including the validated six-item short-form of the Strait Trait Anxiety Inventory (STAI). The STAI is a well-established and validated measure of anxiety that can be used in various clinical settings. The investigators chose the STAI as the primary outcome measure as it has been validated as a measure of anxiety in patients undergoing invasive cardiac procedures. Total score available is 32, minimum score 8. The higher the score the higher the anxiety.

SECONDARY OUTCOMES:
Difference in post procedure satisfaction scores between patients receiving standard care and those who experienced the immersive VR experience | 3 months
  After cardiac catheterisation study patients will be asked to complete a satisfaction questionnaire. This is a modification of an accepted and validated post cardiac catheterisation patient satisfaction questionnaire. Total score available 60. Minimum score 6. Higher score indicates better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Gallagher, MBBS, Principal Investigator — University Hospital of Wales
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No